CLINICAL TRIAL: NCT06901973
Title: Epidemiological, Radiological, Therapeutic and Evolutionary Aspects of Distal Radius Fractures in Adults in South Kivu: a Multi-center Cross-sectional Study.
Brief Title: Distal Radius Fractures in Adults: A Multi-Center Study in South Kivu
Status: Completed | Type: Observational
Sponsor: Official University of Bukavu (Other)
Responsible Party: Sponsor
Other Study IDs: UBukavu
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Distal Radius Fracture
Keywords: DISTAL RADIUS FRACTURES
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intrafocal pinning — Intrafocal pinning involves the percutaneous insertion of Kirschner wires to stabilize the distal radius fracture, often followed by plaster immobilization.

SUMMARY:
The goal of this observational study is to describe the epidemiological, radiological, therapeutic, and evolutionary characteristics of distal radius fractures in adults in the Bukavu Health District, South Kivu, DRC.

. The main question it aims to answer is:

• What are the epidemiological, radiological, therapeutic, and evolutionary characteristics of distal radius fractures in adults in South Kivu, and how does intrafocal nailing influence outcomes such as consolidation time and complication rates in this population?

Participants who have already operated for distal radius fracture will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 17 years or older at the time of injury.
* Diagnosed with a distal radius fracture via clinical and radiological assessment.
* Admitted, treated, and followed up at one of the 16 participating institutions.
* Complete medical records available, including epidemiological, clinical, radiological, therapeutic, and outcome data.

Exclusion Criteria:

* Patients under 17 years of age.

  * Incomplete or missing medical records.
  * Fractures not involving the distal radius.
  * Patients transferred to non-participating facilities without follow-up data.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only male and female
Study Population: The study population consists of adults diagnosed with distal radius fractures (DRFs) who were admitted, treated, and followed up across 16 hospitals and university medical centers in the Bukavu Health District, South Kivu, Eastern Democratic Republic of Congo (DRC), between January 1, 2018, and December 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Time to consolidation | 45 days
  Definition: The duration (in days) from the initiation of treatment with intrafocal pinning to radiological evidence of fracture healing (union), defined as the presence of bridging callus across the fracture site on X-ray.
  Measurement: Calculated retrospectively from medical records, reported as mean ± standard deviation (e.g., 47.56 ± 6.75 days in the study).
  Rationale: Consolidation time is a direct indicator of treatment success, reflecting the intervention's ability to stabilize the fracture and promote healing. It is critical in a resource-limited setting where prolonged recovery impacts patient function and healthcare burden.
  Data Source: Radiology reports and follow-up records.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinics of Bukavu, Bukavu, South Kivu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1. Rundgren J, et al. BMC Musculoskelet Disord. 2020;21(1):88. 2. Chinta SR, et al. J Hand Surg Am. 2024;49(2):123-30. 3. Dworkin M, et al. J Am Acad Orthop Surg Glob Res Rev. 2024;8(4):e23.00282.